CLINICAL TRIAL: NCT04839120
Title: Phase I Clinical Trial of the KLK Inhibitor MDPK67b to Assess Its Pharmacokinetic, Pharmacodynamic, Tolerability and Safety Profile in Healthy Male Volunteers
Brief Title: PK, PD, Tolerability and Safety of MDPK67b in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Med Discovery SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDPK67b-1001
Record Dates: First submitted 2021-03-29; First posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MDPK67b (Active Comparator)
  Interventions: Drug: MDPK67b
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDPK67b — Two subgroups (Panels A and Panel B) of four subjects were to be randomly allocated either to placebo or to three increasing doses of MDPK67b, administered as single infusion at intervals of at least two weeks during the first three periods with the last period involving four repeated doses administered at three-day intervals.
  Arms: MDPK67b
Drug: Placebo — Two subgroups (Panel A and Panel B) of four subjects were to be randomly allocated either to placebo or to three increasing doses of MDPK67b, administered as single infusion at intervals of at least two weeks during the first three periods with the last period involving four repeated doses administered at three-day intervals.
  Arms: Placebo

SUMMARY:
This is a Phase I, single centre, prospective, randomized, alternating panels, ascending doses with interspersed placebo, double-blind, crossover trial.

The trial will include 8 volunteers divided into 2 panels (A and B) investigated in alternance, each submitted to 4 investigation periods following a crossover design in double blind, with ascending intravenous doses of MDPK67b and an interspersed placebo.

The ascending dose sequence ranges from 2 to 48 mg, with 2-fold increase steps (3 to 4- fold increase steps in each individual volunteer). Three single doses will be administered at a minimum of 2 weeks intervals during the first 3 periods, and finally during the last period 4 repeated doses will be administered at a three days intervals, using either the highest dose of the ascending sequence (i.e. 24 or 48 mg) or the maximal tolerated dose (if it has been exceeded in the ascending sequence of single doses).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged between 18 and 45 years
2. Body weight (BW) ranging between 55 and 95 kg, providing body mass index (BMI) is between 18 and 29 kg/m2
3. Absence of significant findings in the medical history and physical examination as judged by the investigator, especially for cardiovascular, pulmonary, haematological and nervous systems
4. Absence of significant laboratory abnormalities as judged by the investigator. Gilbert's syndrome (increased total and unconjugated bilirubin when fasting) will be accepted if mild
5. 12-lead ECG without significant abnormalities
6. Negative urine drug screen (amphetamines, benzodiazepines, cannabis, cocaine, opiates)
7. Negative alcohol breath test
8. Ability to understand the procedures, agreement to participate and willingness to give written informed consent
9. Co-operative attitude and availability for scheduled visits over the entire study period.
10. The subjects will have to refrain from travels outside Europe over the whole study duration.

Exclusion Criteria:

1. History of major cardiovascular, pulmonary, hepatic, immunological, renal, haematological, gastrointestinal, genitourinary, neurological, or rheumatologic disorders
2. Active diseases of any type, including inflammatory disorders and infections. Mild acne is permissible providing no systemic or local treatment is provided or planned (except for cleaning lotions)
3. History of significant allergy or asthma. Allergic rhinitis or conjunctivitis is acceptable if non symptomatic when starting the study and if symptoms are not anticipated to occur during the study to a point that would require corticosteroid therapy (e.g. in case of annual use)
4. History of cardiovascular dysfunction if considered as clinically relevant (conduction abnormality, arrhythmia, bradycardia, angina pectoris, cardiac hypertrophy unless elicited by training, pulmonary embolism)
5. Hypertension defined as supine blood pressure >150/90 mmHg or recurrent hypotensive events considered as clinically relevant or documented orthostatic hypotension
6. Any clinically significant coagulation disorder, based on either clinical manifestations (abnormal bleeding etc.) or abnormal laboratory values (platelet count, TP, aPTT, Thrombin time and fibrinogen).
7. Sick sinus syndrome, known long QT syndrome, reproducible observation of QTc >440 ms or of pronounced sinus bradycardia (<40 bpm)
8. Intense sport activities. Moderate sport is acceptable and activities should remain fairly constant throughout the study
9. Any clinically significant laboratory value on screening that are not within normal range on single repeat (Gilbert's syndrome acceptable if mild)
10. Positive hepatitis B or C antigen screen
11. Positive HIV antibody screen or screen not performed
12. Any recent acute illness or sequelae thereof which could expose the subject to a higher risk or might confound the results of the study
13. Treatment in the previous three months with any drug known to have well-defined potential for toxicity to a major organ
14. History of hypersensitivity to any drug if considered as serious
15. Use of any medication the week prior to study or as based on 5 serum half-life rule and throughout study, including aspirin or other over-the-counter (OTC) preparation. Paracetamol is permissible before and during study as a rescue medication but only with investigator's permission.
16. Participation in a clinical investigation or blood donation of 500 ml within the past 3 months
17. History of relevant alcohol or drug abuse
18. Smoking. Consumption of ≤5 cigarettes/day or equivalent is acceptable providing the subject can refrain from smoking from one week before and during the whole study duration
19. Consumption of a large quantity of coffee, tea, chocolate (more than 4 cups/day) or equivalent (Cola drinks)
20. Present consumption of a large quantity of alcohol or wine (>0.5 L wine/day) or equivalent, (equivalent to more than 35 g ethanol per day).
21. Psychological status which could impact on subject's ability to give informed consent
22. Any feature of subject's medical history or present condition which, in the investigator's opinion, could confound the results of the study, complicate its interpretation, or represent a potential risk for the subject.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | Week 8
  Subjects were assessed for AEs at each visit.
MDPK67b serum level | Up to 144 hours after drug administration
  Serum concentrations of MDPK67b were measured using an ELISA method.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois (CHUV) - Division of Clinical Pharmacology, Lausanne, Switzerland